CLINICAL TRIAL: NCT01513018
Title: Effects of High and Low Tidal Volumes on Arterial Oxygenation and Pulmonary Shunt During One-Lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DEOEC RKEB/IKEB 2976-2009
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Postoperative Lung Injury
Keywords: OLV; one lung ventilation

ARMS (2):
- high (10 ml/kg) tidal volumes (Active Comparator): Evaluate the influence of low (5 ml/kg) and high (10 ml/kg) tidal volumes on arterial oxygenation and Intrapulmonary shunt during one lung ventilation.
  Interventions: Other: high tidal volumes
- low tidal volume (5 ml/kg) (Active Comparator): Evaluate the influence of low (5 ml/kg) and high (10 ml/kg) tidal volumes on arterial oxygenation and Intrapulmonary shunt during one lung ventilation.
  Interventions: Other: low tidal volume

INTERVENTIONS:
Other: high tidal volumes — One-lung ventilation was started at skin incision using a volume-controlled square-wave flow pattern. Patients were randomly assigned to 30 minutes of ventilation with a tidal volume of 10 ml/kg tidal volume without external PEEP and respiratory rate of 10 breaths/minute (n=50) or to a tidal volume of 5 ml/kg with 5 cmH2O PEEP and a respiratory rate of 20 breaths/minute (n=50). Minute volume was thus kept constant during each experimental condition.
  Randomization was based on computer-generated codes that were maintained in sequentially numbered sealed opaque envelopes until after induction of anesthesia. During the subsequent 30 minutes of one-lung ventilation, the alternative ventilatory management was used.
  Arms: high (10 ml/kg) tidal volumes
Other: low tidal volume — One-lung ventilation was started at skin incision using a volume-controlled square-wave flow pattern. Patients were randomly assigned to 30 minutes of ventilation with a tidal volume of 10 ml/kg tidal volume without external PEEP and respiratory rate of 10 breaths/minute (n=50) or to a tidal volume of 5 ml/kg with 5 cmH2O PEEP and a respiratory rate of 20 breaths/minute (n=50). Minute volume was thus kept constant during each experimental condition.
  Randomization was based on computer-generated codes that were maintained in sequentially numbered sealed opaque envelopes until after induction of anesthesia. During the subsequent 30 minutes of one-lung ventilation, the alternative ventilatory management was used.
  Arms: low tidal volume (5 ml/kg)

SUMMARY:
The ideal tidal volume (TV) during one-lung ventilation (OLV) remains controversial. High tidal volumes may increase the incidence of postoperative lung injury after thoracic surgery. The investigators thus evaluated the influence of low (5 ml/kg) and high (10 ml/kg) tidal volumes on arterial oxygenation and Intrapulmonary shunt during OLV.

One hundred patients scheduled for thoracic surgery were enrolled. During OLV, patients were randomly assigned to 30 minutes of ventilation with high TV (10 ml/kg with zero end-expiratory pressure (ZEEP)) at a rate of 10 breaths/minute or low tidal volume (5 ml/kg with 5 cm H2O positive end-expiratory pressure (PEEP)) at a rate of 20 breaths/minute. During the subsequent 30 minutes, each patient received the alternative management. Minute volume was thus kept constant during each experimental condition. Arterial blood partial pressures, hemodynamic responses, and ventilatory parameters were recorded. Results are presented as means ± SDs; P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III patients scheduled for lung resection surgery.

Exclusion Criteria:

* severe cardiovascular disease
* severe alteration of the preoperative pulmonary function, with FEV1 70-120% predicted and FEV1/FVC ≥ 70% predicted considered to be normal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
low (5ml/kg) tidal volume on arterial oxygenation | 30 minutes of ventillation
  Evaluate the influence of low (5 ml/kg) and high (10 ml/kg) tidal volumes on arterial oxygenation and Intrapulmonary shunt during one lung ventilation.
high (10 ml/kg) tidal volumes on arterial oxygenation | 30 minutes of ventillation
  Evaluate the influence of low (5 ml/kg) and high (10 ml/kg) tidal volumes on arterial oxygenation and Intrapulmonary shunt during one lung ventilation.
low (5 ml/kg)tidal volumes on Intrapulmonary shunt | 30 minutes of ventillation
  Evaluate the influence of low (5 ml/kg) and high (10 ml/kg) tidal volumes on arterial oxygenation and Intrapulmonary shunt during one lung ventilation.
high (10 ml/kg) tidal volumes on Intrapulmonary shunt | 30 minutes of ventillation
  Evaluate the influence of low (5 ml/kg) and high (10 ml/kg) tidal volumes on arterial oxygenation and Intrapulmonary shunt during one lung ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Tamás Végh, M.D., Principal Investigator — Klinikum Ludwigshafen
Locations (1):
- University of Debrecen, Medical and Health Science CenterDepartment of Anesthesiology and Intensive Care, Debrecen, Hungary